CLINICAL TRIAL: NCT01025271
Title: Cerebrospinal Fluid Pharmacokinetics of Daptomycin
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: unable to enroll subjects study stopped due to lack of enrollment
Sponsor: University of Pittsburgh (Other)
Collaborators: Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB#: PRO09070202
Record Dates: First submitted 2009-12-02; First posted 2009-12-03 (Estimated); Results first posted 2013-08-12 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2013-08

CONDITIONS: Meningitis
Keywords: meningitis
MeSH Terms: conditions — Meningitis | interventions — Daptomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- open label (Other): patients meeting entry criteria enrolled and pk samples obtained around dosing of daptomycin
  Interventions: Drug: Daptomycin

INTERVENTIONS:
Drug: Daptomycin — one dose of daptomycin (10 milligrams of the drug per kilogram of the subject's body weight

SUMMARY:
This is a prospective pharmacokinetic study in patients having external ventricular drains with suspected external ventricular drain related bacterial meningitis. A single dose of daptomycin will be administered for the purposes of the study and PK samples will be obtained around this dosing.

DETAILED DESCRIPTION:
information related to the subject's demographics, past medical history and current medical history will be collected from the medical record. This will be collected by the research coordinator.

The following samples will be obtained by the research coordinator or bedside RN and sent to UPMC laboratory for evaluation.

1 teaspoon of blood for creatinine phosphokinase level will be obtained

pregnancy testing will occur if necessary - 1 teaspoon of blood Screening procedures about 30 minutes of the patient's time includes, medical record review will occur and information related to the patients past medical history, demographics, and present condition, results of present testing will be collected, pregnancy test- 1 teaspoon of blood, creatinine phosphokinase - 1 teaspoon of blood. Additionally another CPK level will be obtained 36 hours post daptomycin infusion. This blood sample is a routine part of your clinical care. The bedside RN or research coordinator will collect the blood samples and send to the lab at UPMC for evaluation and the medical chart review will be completed by research coordinator.

if the patient meets entry criteria the following will occur at the patient's bedside in their room. If there is a clinical indication that requires the catheter to be removed, the removal will not be delayed for the purposes of the research study:

Patient will receive one dose of daptomycin via IV given by the bedside RN over 30 minutes (the dosing will be based on the patient's weight- 10 milligrams per kilogram). PK sampling will be obtained around this dosing. 10 PK samples around dosing of Daptomycin will occur- this will be approximately 11 teaspoons (1 teaspoon per sample) and will be obtained immediately before the Daptomycin dosing, then 1, 2, 4, 8, 10, 16, 24 and 36 hours after the end of infusion. The research coordinator will come to the bedside and the bedside RN will obtain these samples and will be obtained via the patient's existing IV catheter or central line.

4 samples of cerebrospinal fluid approximately 1 teaspoon per sample will be collected on the day daptomycin is given. These samples will be obtained by the bedside RN and taken from the already existing spinal fluid draining catheter.

10 subjects will have these samples obtained 1, 8, 16, 24 after the end of the daptomycin infusion and 10 subjects will have them collected at 2,4, 10 and 36 hours after the end of the daptomycin infusion.

2 days after collection of PK samples the patient will be seen at their bedside to check how well the patient is doing. This will take 5-10 minutes of the patient's time. If the patient is d/c home a research coordinator will call the patient to check on their status again this will take about 5-10 minutes

ELIGIBILITY:
Inclusion Criteria:

Adults with suspected EVD related meningitis or ventriculitis who already have an external ventricular drain placed, as part of standard clinical care for CSF drainage, and whose clinicians plan to start antibiotics. There should be a clinical indication for the EVD to be in place for ≥ 72 hrs. An intravenous line which can be accessed for blood draws should be present.

Exclusion Criteria:

Age less than 18 years of age Patient is a woman who is pregnant or lactating Allergies or prior adverse reactions to daptomycin, which would preclude its use.

Elevated CK levels (>500). Inability to obtain informed consent or get proxy consent. Patients on CRRT (continuous renal replacement therapies) or on dialysis Patients with an estimated CrCl <30 cc/min as estimated by MDRD at base line. Patients with a BMI >30 Any medical condition leading to a life expectancy of < 48 hours, as determined by the clinician.

Patient who have received a dose of daptomycin in the last 7 days. Patients is participating in other studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2010-05; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karin Byers, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: unable to meet enrollment no data available. Study terminated early
Pre-assignment Details: unable to meet enrollment no data available. Study terminated early
Period: Overall Study
Arm/Group | Open Label
Started | 2 (unable to meet enrollment no data available. Study terminated early)
Completed | 2 (unable to meet enrollment no data available. Study terminated early)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Open Label
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Characterize the CSF and Plasma Concentration-time Profile of Daptomycin in Patients With External Ventricular Drain (EVD) Related Meningitis
Description: unable to meet enrollment no data available. Study terminated early
Time Frame: 5 years
Population: unable to meet enrollment no data available. Study terminated early
Arm/Group | Open Label
Number analyzed (Participants) | 0

2. Secondary Outcome: Characterize the CSF and Plasma Concentration-time Profile of Daptomycin in Patients With External Ventricular Drain (EVD) to Determine the CSF Penetration and Pharmacokinetic Parameters in This Patient Population (
Description: no analysis completed
Time Frame: 5 years
Groups:
- PK Sampling: patients meeting entry criteria enrolled and pk samples obtained around dosing of daptomycin
Arm/Group | PK Sampling
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Open Label
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

LIMITATIONS AND CAVEATS:
unable to meet enrollment no data available.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No